CLINICAL TRIAL: NCT02947659
Title: The Relationship Between the Development of Musculoskeletal Disorders and Body Mass Index and Academic Stress in Bahraini University Students
Brief Title: Body Mass Index, Academic Stress and Musculoskeletal Disorders Relationships
Status: Completed | Type: Observational
Sponsor: Ahlia University (Other)
Responsible Party: Principal Investigator, Dr Sayed Tantawy, Associate Professor of Physiotherapy, Ahlia University
Other Study IDs: 2015/16001
Record Dates: First submitted 2016-10-18; First posted 2016-10-28 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: BMI, Academic Stress and MSDs Relationships
Keywords: Body mass index; Academic stress; Musculoskeletal disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
[Purpose] To investigate the prevalence of musculoskeletal disorders among healthy students of Ahlia University and to determine the relationship between the prevalence of musculoskeletal disorders and academic stressors and body mass index. [Subjects and Methods]: Self-administered questionnaires were distributed to 94 students aged 18-26 years who were enrolled at various Ahlia University colleges and met other inclusion criteria. The students responded to the standardized Nordic musculoskeletal questionnaire and the modified College Student Stress Inventory regarding musculoskeletal symptoms and academic stressors. Height and weight measurements were also obtained to determine body mass index.

Keywords: Body mass index, Academic stress, Musculoskeletal disorders

DETAILED DESCRIPTION:
[Purpose] To investigate the prevalence of musculoskeletal disorders among healthy students of Ahlia University and to determine the relationship between the prevalence of musculoskeletal disorders and academic stressors and body mass index. [Subjects and Methods]: Self-administered questionnaires were distributed to 94 students aged 18-26 years who were enrolled at various Ahlia University colleges and met other inclusion criteria. The students responded to the standardized Nordic musculoskeletal questionnaire and the modified College Student Stress Inventory regarding musculoskeletal symptoms and academic stressors. Height and weight measurements were also obtained to determine body mass index.

Keywords: Body mass index, Academic stress, Musculoskeletal disorders

ELIGIBILITY:
Inclusion Criteria:

* A total of 28 male and 66 female students (age, 18-26 years; mean, 21 ± 1.9 years) from various Ahlia University colleges were recruited to participate in this study.
* To be included in the study, all subjects had to be enrolled in an undergraduate program at Ahlia University, Bahrain.
* In addition, they had to be relatively healthy with no diagnosed medical conditions that would cause pain.

Exclusion Criteria:

* Exclusion criteria were previous injury or trauma to body parts, any surgical intervention, history of psychological disorders prior to enrolment at the university, and severe physical disability causing pain.
* In addition, students with blood disorders, such as sickle cell anaemia and thalassaemia, were excluded.

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: A total of 28 male and 66 female students (age, 18-26 years; mean, 21 ± 1.9 years) from various Ahlia University colleges were recruited to participate in this study.
Sampling Method: Probability Sample
Enrollment: 94 (Actual)
Dates: Start 2015-10; Primary Completion 2016-03 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
BMI and MSDs relationship | 10 months

SECONDARY OUTCOMES:
BMI and Academic Stress Relationship | 10 months